CLINICAL TRIAL: NCT07027943
Title: Evaluation Of The Diamine Oxidase Supplementation Effect In Patients With Insomnia Symptoms
Acronym: DAO-SLEEP-2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotek (Industry)
Collaborators: AdSalutem Sleep Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DAO-SLEEP-2023
Record Dates: First submitted 2025-06-06; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Insomnia; Insomnia Type; Sleep Disorder
Keywords: insomnia; diamine oxidase (DAO); DAO supplementation; double-blind; placebo-controlled
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DAO; once per day (Experimental): Gastro-resistant DAO tablets of porcine kidney protein extract. Posology: 3 tablets per day (total 12.6mg of DAO extract/day); once per day.
  Interventions: Dietary Supplement: DAO supplement
- Placebo; once per day (Placebo Comparator): Tablets containing microcrystalline cellulose and hydroxypropyl cellulose, with the same shape, size, and color as the DAO-containing tablets.
  Posology: 3 tablets per day, once per day.
  Interventions: Dietary Supplement: Placebo
- DAO; 3 times per day (Experimental): Gastro-resistant DAO tablets of porcine kidney protein extract. Posology: 3 tablets per day (total 12.6mg of DAO extract/day) in 3 different times per day.
  Interventions: Dietary Supplement: DAO supplement
- Placebo, 3 times per day (Placebo Comparator): Tablets containing microcrystalline cellulose and hydroxypropyl cellulose, with the same shape, size, and color as the DAO-containing tablets. Posology: 3 tablets per day in 3 different times per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DAO supplement — Gastro-resistant DAO tablets of porcine kidney protein extract. Posology: 3 tablets per day (total 12.6mg of DAO extract/day).
  Arms: DAO; 3 times per day; DAO; once per day
Dietary Supplement: Placebo — Tablets containing microcrystalline cellulose and hydroxypropyl cellulose, with the same shape, size, and color as the DAO-containing tablets. Posology: 3 tablets per day.
  Arms: Placebo, 3 times per day; Placebo; once per day

SUMMARY:
Considering the high prevalence of DAO enzyme deficiency in patients referring insomnia symptoms, it would be plausible that the appearance of insomnia symptoms were explained by the DAO enzyme deficiency.

One of the strategies to revert DAO enzyme deficiency would be to supplement patients with DAO enzyme, helping at recovering the normal DAO levels. Therefore, the objective of the present study is to evaluate the effect of DAO enzyme supplementation on the insomnia symptoms characteristics in patients with insomnia symptoms and genetic DAO deficiency as expected from bearing at least one of the 4 above-mentioned SNPs of the AOC1 gene.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* With the ability to understand and sign informed consent reviewed and approved by the Grupo Hospitalario Quironsalud-Catalunya.
* That refer one or more symptoms of insomnia, these being: Difficulty initiating sleep, Difficulty maintaining sleep, Waking up early with inability to go back to sleep.
* Who are carriers, either heterozygous or homozygous, of at least one of the following 4 SNPs associated with a reduction in the enzymatic activity of DAO or a decreased transcriptional activity of it: c.47C>T (rs10156191), c.995C>T (rs1049742), c.1990C>G (rs1049793), c.-691G>T (rs2052129).
* With the ability to attend the foreseen face-to-face and telephonic study visits.
* With the ability to intake the product under study
* Explicit agreement on study participation by reading, understanding, and signing the informed consent reviewed and approved by the Grupo Hospitalario Quironsalud-Catalunya

Exclusion Criteria:

* Insomnia symptoms referred by patients that might be explained by other co-morbid sleep disorders, e.g., narcolepsy, circadian rhythm disturbances, parasomnia, etc.
* Taking DAO supplementation less than 1 month prior to the start of the study.
* Following a diet low in histamine less than 1 month prior to the start of the study.
* Volunteers with allergies to some of the ingredients of the product under study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).

SECONDARY OUTCOMES:
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the SNP variants of AOC1 gene. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the use of insomnia pharmacological treatment (benzodiazepines, melatonin, others, or no pharmacological treatment). Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the SNP variants of AOC1 gene. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the SNP variants of AOC1 gene. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Pittsburgh Sleep Quality Index (PSQI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the use of insomnia pharmacological treatment (benzodiazepines, melatonin, others, or no pharmacological treatment). Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Pittsburgh Sleep Quality Index (PSQI) scale after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions in the Pittsburgh Sleep Quality Index (PSQI) scale after one month of DAO supplementation, compared to the placebo group, stratified by the SNP variants of AOC1 gene. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who reduce at least one point on Component 2 (Sleep latency) of the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who reduce at least one point on Component 2 (Sleep latency) of the Pittsburgh Sleep Quality Index (PSQI) scale, after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who reduce at least one point on Component 5 (Sleep disturbance) of the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who reduce at least one point on Component 5 (Sleep disturbance) of the Pittsburgh Sleep Quality Index (PSQI) scale, after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Number (absolute and percentage) of patients who reduce at least one point on Component 7 (Daytime dysfunction) of the Pittsburgh Sleep Quality Index (PSQI) scale | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who reduce at least one point on Component 7 (Daytime dysfunction) of the Pittsburgh Sleep Quality Index (PSQI) scale, after one month of DAO supplementation, compared to the placebo group. Score goes from 0 to 21. A higher score indicates a worse outcome in sleep quality.
Serum DAO activity levels | Visit day 0 and day 28.
  Mean increase of serum DAO activity levels after one month of DAO supplementation, compared to the placebo group.
Number (absolute and percentage) of patients who increase their serum DAO activity levels | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who increase their serum DAO activity levels after one month of DAO supplementation, compared to the placebo group
Mean DAO baseline activity levels | Visit day 0 and day 28.
  Mean DAO baseline activity levels stratified by the SNP variants of AOC1 gene.
Mean increase in DAO activity levels | Visit day 0 and day 28.
  Mean increase in DAO activity levels, after one month of DAO supplementation, compared to the placebo group, stratified by the SNP variants of AOC1 gene.
Number (absolute and percentage) of patients who improve their symptoms associated with histamine intolerance due to DAO deficiency | Visit day 0 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms associated with histamine intolerance due to DAO deficiency, after one month of DAO supplementation, compared to the placebo group.
Number (absolute and percentage) of patients who refer improvement in their daytime repercussions of insomnia | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who refer improvement in their daytime repercussions of insomnia (such as drowsiness, fatigue, cognitive deficit, lack of concentration, lack of attention or memory, mood swings, and/or headaches) after one month of DAO supplementation, compared to the placebo group.
Number (absolute and percentage) of patients in the once-a day groups who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients in the once-a day groups who improve their symptoms of insomnia and daytime repercussions by at least one point in the ISI scale after one month of DAO supplementation compared to placebo. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Percentage of doses taken of DAO supplementation | Visit day 0 and day 28.
  Percentage of doses taken of DAO supplementation over one month period (counting leftover medication and with patient interview) in the once-a-day groups compared to placebo.
Number (absolute and percentage) of patients in the three times per day groups who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients in the three times per day groups who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation compared to placebo. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Percentage of doses taken of DAO supplementation | Visit day 0 and day 28.
  Percentage of doses taken of DAO supplementation over one month period (counting leftover medication and with patient interview) in the three times per day groups compared to placebo
Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale | Visit day 0, day 7, day 14, day 21 and day 28.
  Number (absolute and percentage) of patients who improve their symptoms of insomnia and daytime repercussions by at least one point in the Insomnia Severity Index (ISI) scale after one month of DAO supplementation in the once-a-day group compared to the three times per day group. Score goes from 0 to 28. A higher score indicates a worse outcome (severity of insomnia).
Percentage of doses taken of DAO supplementation | Visit day 0 and day 28.
  Percentage of doses taken of DAO supplementation over one month period (counting leftover medication and with patient interview) in the once-a-day groups compared to three times per day.
Percentage of compliant patients | Visit day 0 and day 28.
  Percentage of compliant patients (compliance percentage > 80%) over one month period (counting leftover medication and with patient interview) in the once-a-day groups compared to placebo.
Percentage of compliant patients | Visit day 0 and day 28.
  Percentage of compliant patients (compliance percentage > 80%) over one month period (counting leftover medication and with patient interview) in the three times per day groups compared to placebo.
Percentage of doses taken of DAO supplementation | Visit day 0 and day 28.
  Percentage of doses taken of DAO supplementation over one month period (counting leftover medication and with patient interview) in the once-a-day group compared with the three times per day group.
Percentage of compliant patients | Visit day 0 and day 28.
  Percentage of compliant patients (compliance percentage > 80%) over one month period (counting leftover medication and with patient interview) in the once-a-day group compared with the three times per day group.
Report of adverse events | Visit day 0, day 7, day 14, day 21 and day 28.
  Report of adverse events after one month of DAO supplementation, compared to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Karol Enrique Uscamaita Amaut, MD, Principal Investigator — AdSalutem Sleep Institute
Locations (1):
- AdSalutem Sleep Institute, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
ISI score and PSQI score
Supporting Information: Study Protocol
Time Frame: According to legislation

REFERENCES:
- [Derived] Ferrer-Garcia J, Navarro MD, Abadias M, Lopez-Garcia R, Sansalvador A, Gris G, Uscamaita K. Effect of diamine oxidase (DAO) enzyme dietary supplementation in subjects with insomnia symptoms and single nucleotide polymorphisms of the AOC1 gene: a randomized double-blind placebo-controlled study. Sleep Med X. 2025 Dec 1;11:100167. doi: 10.1016/j.sleepx.2025.100167. eCollection 2026 Dec. PMID 41437955